CLINICAL TRIAL: NCT06698926
Title: A Phase 1 First in Human, Single and Multiple Ascending Dose, Food Effect, and Drug-Drug Interaction Study in Healthy Volunteers to Evaluate the Safety, Tolerability, and Pharmacokinetics of ABBV-CLS-616
Brief Title: A Study to Assess the Safety, Tolerability, and Interactions of ABBV-CLS-616 Oral Tablets in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Calico Life Sciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: M25-206
Record Dates: First submitted 2024-11-06; First posted 2024-11-21 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-CLS-616
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (14):
- Part 1: Group 1 (Experimental): Participants will receive either ABBV-CLS-616 Dose A or placebo after fasting on Day 1 and will be confined for 19 days.
  Interventions: Drug: ABBV-CLS-616; Drug: Placebo
- Part 1: Group 2 (Experimental): Participants will receive either ABBV-CLS-616 Dose B or placebo after fasting on Day 1 and will be confined for 19 days.
  Interventions: Drug: ABBV-CLS-616; Drug: Placebo
- Part 1: Group 3 (Experimental): Participants will receive either ABBV-CLS-616 Dose C or placebo after fasting on Day 1 and will be confined for 8 days.
  Interventions: Drug: ABBV-CLS-616; Drug: Placebo
- Part 1: Group 4 (Experimental): Participants will receive either ABBV-CLS-616 Dose D or placebo after fasting on Day 1 and will be confined for 8 days.
  Interventions: Drug: ABBV-CLS-616; Drug: Placebo
- Part 1: Group 5 (Experimental): Participants will receive either ABBV-CLS-616 Dose E or placebo after fasting on Day 1 and will be confined for 8 days.
  Interventions: Drug: ABBV-CLS-616; Drug: Placebo
- Part 1: Group 6 (Experimental): Participants will receive either ABBV-CLS-616 Dose F or placebo after fasting on Day 1 and will be confined for 8 days.
  Interventions: Drug: ABBV-CLS-616; Drug: Placebo
- Part 2: Group 7 (Experimental): Participants will receive either ABBV-CLS-616 Dose G or placebo daily, starting on Day 1 for 7 days and will be confined for 14 days.
  Interventions: Drug: ABBV-CLS-616; Drug: Placebo
- Part 2: Group 8 (Experimental): Participants will receive either ABBV-CLS-616 Dose H or placebo daily, starting on Day 1 for 7 days and will be confined for 14 days.
  Interventions: Drug: ABBV-CLS-616; Drug: Placebo
- Part 2: Group 9 (Experimental): Participants will receive either ABBV-CLS-616 Dose D or placebo daily, starting on Day 1 for 7 days and will be confined for 14 days.
  Interventions: Drug: ABBV-CLS-616; Drug: Placebo
- Part 2: Group 10 (Experimental): Participants will receive either ABBV-CLS-616 Dose E or placebo daily, starting on Day 1 for 7 days and will be confined for 14 days.
  Interventions: Drug: ABBV-CLS-616; Drug: Placebo
- Part 2: Group 11 (Experimental): Participants will receive either ABBV-CLS-616 Dose F or placebo daily, starting on Day 1 for 7 days and will be confined for 14 days.
  Interventions: Drug: ABBV-CLS-616; Drug: Placebo
- Part 3: Sequence 1 (Experimental): In Period 1, participants will receive ABBV-CLS-616 Dose C on Day 1 after fasting and will be confined for 7 days. In Period 2, participants will receive ABBV-CLS-616 Dose C on Day 1, without fasting and will be confined for 8 days.
  Interventions: Drug: ABBV-CLS-616
- Part 3: Sequence 2 (Experimental): In Period 1, participants will receive ABBV-CLS-616 Dose C on Day 1 without fasting and will be confined for 7 days. In Period 2, participants will receive ABBV-CLS-616 Dose C on Day 1, after fasting and will be confined for 8 days.
  Interventions: Drug: ABBV-CLS-616
- Part 4: Itraconazole (Experimental): In Period 1, participants will receive ABBV-CLS-616 Dose C on Day 1, after fasting and will be confined for 7 days. In Period 2, participants will receive Itraconazole daily for 10 days without fasting and will receive ABBV-CLS-616 Dose C on Day 4 after fasting. Participants will be confined for 11 days.
  Interventions: Drug: ABBV-CLS-616; Drug: Itraconazole

INTERVENTIONS:
Drug: ABBV-CLS-616 — Oral Tablet
Drug: Placebo — Oral Tablet
  Arms: Part 1: Group 1; Part 1: Group 2; Part 1: Group 3; Part 1: Group 4; Part 1: Group 5; Part 1: Group 6; Part 2: Group 10; Part 2: Group 11; Part 2: Group 7; Part 2: Group 8; Part 2: Group 9
Drug: Itraconazole — Oral Capsule
  Arms: Part 4: Itraconazole

SUMMARY:
This is a Phase 1, first in human, randomized, four-part study to investigate the safety, tolerability, and pharmacokinetics of ABBV-CLS-616 after oral dosing in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Part 2 only: Participant must have normal platelet count at screening and upon initial confinement.
* Part 2 only: Participant must not have known or suspected coagulopathy, or prothrombin time (PT)/activated partial thromboplastin time (aPTT)/international normalized ratio (INR) values outside of normal range at screening.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, neurological examination, ophthalmic examination (Part 2 only) laboratory profile and a 12-lead Electrocardiogram.

Exclusion Criteria:

* Part 2 only: Clinically significant active or recurrent ocular disease.
* Part 2 only: History of lumbar puncture and/or collection of cerebrospinal fluid within 30 days prior to Screening.
* Part 2 only: History of current condition of chronic lower back pain.
* Evidence of conditions that might preclude the subject from undergoing a lumbar puncture.
* History of clinically significant neurological epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, coagulopathy, or any uncontrolled medical illness.
* History of suicidal ideation within one year prior to study drug administration as evidenced by answering "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia Suicide Severity Rating Scale completed at Screening, or any history of suicide attempts within the last two years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to approximately 90 days
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 270532, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-206